CLINICAL TRIAL: NCT00422955
Title: A 16-week, Randomised, Double-blind, Placebo-controlled, Single-centre Study to Investigate Fluid Retention in Insulin-treated Subjects With Type 2 Diabetes Mellitus and Varying Degrees of Autonomic Neuropathy When Administered Rosiglitazone 4mg Twice Daily
Brief Title: Fluid Retention in Rosiglitazone Treated Subjects With Autonomic Neuropathy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 49653/376
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Neuropathy, Diabetic
Keywords: fluid retention; Autonomic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
Fluid management study in patients with type 2 diabetes and autonomic neuropathy.

ELIGIBILITY:
Inclusion criteria:

* Subjects with Type 2 Diabetes (T2DM) as defined by the 1999 WHO criteria [World Health Organisation , 1988/NCD/NCS/99.2] with stable FPG of = 7.0 and = 15.0 mmol/l who have been established on insulin therapy for at least 6 months
* BMI = 40 kg.m2
* Subject who is willing and able to provide a signed and dated written informed consent.

Exclusion Criteria:

* Subjects with an HbA1c level > 12%
* Subjects taking oral hypoglycaemic agents other than metformin
* Subjects on insulin dosage > 200 units/day

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-11; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change in transcapillary escape rate of L125 albumin following 16 weeks treatment

SECONDARY OUTCOMES:
Change in plasma volume, pedal oedema, extracellular fluid volume following 16 weeks treatment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Rennings AJ, Smits P, Stewart MW, Tack CJ. Autonomic neuropathy predisposes to rosiglitazone-induced vascular leakage in insulin-treated patients with type 2 diabetes: a randomised, controlled trial on thiazolidinedione-induced vascular leakage. Diabetologia. 2010 Sep;53(9):1856-66. doi: 10.1007/s00125-010-1787-8. Epub 2010 May 25. PMID 20499046
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 49653/376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 49653/376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 49653/376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 49653/376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 49653/376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 49653/376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register